CLINICAL TRIAL: NCT02563275
Title: The Operation of Control Devices During Parabolic Flights: Influence of Weightlessness, Stress and Motivation
Acronym: Grafism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-002
Record Dates: First submitted 2015-07-22; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human fine motor skills measurements during weightlessness (Other)
  Interventions: Other: motion analysis system; Other: parabolic flight

INTERVENTIONS:
Other: motion analysis system
Other: parabolic flight

SUMMARY:
The aim of this project is to investigate whether alterations in sensory-motor performances during weightlessness are only of theoretical relevance, or indeed restrict the capacity of the participants. To find out, volunteers will monitor a complex realistic process by operation of buttons and switches in weightlessness. The task will mimic the control of vehicles, research equipment and industrial processes. Effects of weightlessness will be separated from effects induced by stress and those of motivation through evaluation of cortisol and manipulation of motivation.

DETAILED DESCRIPTION:
Investigations description

---------------------------------- Subjects will sit in a rack at a table in front of a 17" screen of an Eye Tracker system (Tobii® T60). The right part of the screen will be covered by a row of operating devices; two rotary knobs of different size, one turn switch and one simple push button. The construction of these devices is based on real ones on board the ISS. Integrated in three of these devices are force sensors (6D ATI® Nano17), which register grip torques and forces while subjects' manipulate the devices.

Four Vicon® Bonita cameras are positioned over the table and attached to a table-fixed metal frame. They will register hand dynamics throughout all grasping movements in normal gravity as well as in microgravity.

In accordance to a classical control task by Kramer (1999) subjects will be asked to control pointer instruments, which are displayed one below the other on the screen. These controls will be embedded in a real life scenario where subjects have to react on specific signals within this scenario: As soon as one of the displayed pointers reach a critical deflection, subjects have to react as fast as possible by grasping towards the associated control device, rotate or push it and turn back to the starting position. This action will bring the pointers back to an uncritical position. The pointers will move independent from the others. Additionally we introduce one compatible and one incompatible pointer-device connection, i.e. the upper pointer can be controlled with the lower device, the middle pointer with the middle and the lower pointer with the upper device.

Equipment used --------------------- Hand movements Hand movements are registered from above and the side by four infrared high-speed cameras (Bonita Vicon-Cameras - CE mark 0088) which register with 250Hz the 3D positions of ten small reflexive markers (attached by double sided adhesive tape to all fingertips and to the thumb of the subjects' right hand). The cameras are connected via cables with an Ultranet which is the central processing unit. The Ultranet is connected with a network cable to a corresponding desktop computer.

Force and torque sensors The different knobs (three of them) that have to be grasped, measure forces and torques applied to it at a rate of 250Hz. These sensors (Nano 17 of the ATI DAQ F/T System) are connected to power supply boxes with a booster, which supplies the data via a DAQ card to the desktop computer. We will analyze usual force parameters such as initial forces at the knob, but also maximal forces applied to the knobs.

Experimental protocol

----------------------------- Before flight subjects will be familiarized with the setup and the protocol. For each flight day, only one subject will be studied. The procedure will be the same on each flight.

Overall one subject will be tested during 26 parabolas. Within the first 13 parabolas motivational state will be manipulated in a positive way by means of positive word presentation (subliminal priming) and within the last 13 parabolas with negative words. The order of positive versus negative priming will be counterbalanced across subjects.

All subjects perform the task of operating control devices once in level flight before the first parabolas, during the parabolas and after the parabolas. After the whole flight subjects will perform the control task again.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 21 to 65
* Right handed
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude .There will be no additional test performed for subject selection.

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Person with medical history of neurological disorders
* Person with medical history of musculoskeletal disorders of the lower limbs, especially of the ankle and knee joint.
* Pregnant women

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Velocity (deg/sec) of the right hand movement measured with a motion analysis system | baseline
Forces (Newton) applied by the hand on the objects to be grasped measured with strain gauges | baseline
Torques (N.m) applied by the hand on the objects to be grasped measured with strain gauges | baseline
Peak velocity (deg/sec) of the right hand measured with a motin analysis system | baseline
Initial force (Newton) on the grasped object measured with strain gauges | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France